CLINICAL TRIAL: NCT01204385
Title: Identification and Characterization of the Bacteria Causing Acute Otitis Media (AOM) Episodes in Young Children in Saudi Arabia
Brief Title: Study to Identify and Characterize the Bacteria Causing Acute Otitis Media Episodes in Young Children in Saudi Arabia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111337
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Infections, Streptococcal
Keywords: Non-typeable Haemophilus Influenzae; Acute Otitis Media; Streptococcus Pneumoniae; etiology
MeSH Terms: conditions — Streptococcal Infections; Otitis Media | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Middle ear fluid and urine

GROUPS / COHORTS (1):
- Study Group
  Interventions: Procedure: Sample collection

INTERVENTIONS:
Procedure: Sample collection — Middle ear fluid and urine

SUMMARY:
The purpose of the study is to identify the bacterial aetiology of acute otitis media episodes in young children aged ≥ 3 months to < 5 years in Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

A child will be eligible for inclusion if he/she meets the following criteria:

* Age: ≥ 3 months and < 5 years at the time of enrolment. The subject becomes ineligible on the fifth birthday.
* Signs, symptoms, and conditions: i. One of the functional or general signs of otalgia (or its equivalent: irritability), conjunctivitis, fever AND EITHER ii. Paradise's criteria (bulging, diffused or localised inflamed tympanic membranes) OR iii. Spontaneous otorrhoea of less than 24 hours
* Onset of signs and symptoms of AOM within 72 hours prior to diagnosis of AOM by a physician. To be included as treatment failure, subjects must have then received antibiotic treatment from the physician, but remain symptomatic 48-72h after initiation of treatment
* Written informed consent obtained from parent or guardian prior to study start.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply, the child must not be included in the study.

* Hospitalised during the diagnosis of AOM or during treatment,
* Otitis externa, or otitis media with effusion
* Presence of a transtympanic aerator
* Systemic antibiotic treatment received for a disease other than AOM in the 72 hours prior to enrolment,
* Receiving antimicrobial prophylaxis for recurrent AOM,
* Provision of antibiotic by paediatrician/ENT specialist at the enrolment visit, prior to the sampling
* Patients on antibiotics for AOM who are clinically improving.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects aged ≥ 3 months and < 5 years of age, diagnosed as having AOM
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of H. influenzae, S. pneumoniae and other bacterial pathogens isolated from middle ear fluid samples | Average time frame: 12 months

SECONDARY OUTCOMES:
Occurence of H. influenzae and S. pneumoniae serotypes | Average time frame: 12 months
Antimicrobial susceptibility of H. influenzae, S. pneumoniae and Moraxella catarrhalis isolated from middle ear fluid samples as assessed by standard microbiological techniques | Average time frame: 12 months
Occurrence of treatment failure of acute otitis media and of recurrent acute otitis media (≥ 3 episodes in the last 6 months or ≥ 4 episodes in 12 months) | Average time frame: 12 months
Occurrence of spontaneous otorrhea | Average time frame: 12 months
Occurrence of H. influenzae in acute otitis media cases with treatment failure and in new acute otitis media cases without treatment therapy | Average time frame: 12 months
Occurrence of H. influenzae in acute otitis media cases vaccinated with a pneumococcal vaccine | Average time frame: 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Riyadh, Saudi Arabia